CLINICAL TRIAL: NCT01165762
Title: Total Lymphoid Irradiation, Anti-Thymocyte Globulin and Purified Donor CD34+ and T-cell Transfusion in HLA Haplotype Match Living Donor Kidney Transplantation
Brief Title: Combined Blood Stem Cell and Kidney Transplant of One Haplotype Match Living Donor Pairs.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Everett Meyer (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Everett Meyer, Associate Professor of Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SU-06232010-6408; P01HL075462 (NIH)
Record Dates: First submitted 2010-07-13; First posted 2010-07-20 (Estimated); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: ESRD
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Immune Tolerance; Kidney Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Immune Tolerance, Kidney transplantation (Experimental): Induction of immune tolerance in Haplotype matched living donor kidney transplantation.
  Interventions: Drug: Immune Tolerance

INTERVENTIONS:
Drug: Immune Tolerance — Immune tolerance Kidney and hematopoietic cell transplantation with a conditioning regimen of total lymphoid irradiation and antithymocyte globulin followed by immunosuppressive drugs for 18 months. Immunosuppressive drugs are stopped if stable chimerism is achieved and there is no rejection of the transplant kidney.
  The IDE used in this study is the column used for hematopoietic cell sorting.
  Other Names: Kidney transplantation

SUMMARY:
The Stanford Medical Center Program in Multi-Organ Transplantation and the Division of Bone marrow Transplantation are enrolling patients into a research study to determine if donor stem cells given after a living related one Haplotype match kidney transplantation will change the immune system such that immunosuppressive drugs can be completely withdrawn.

DETAILED DESCRIPTION:
The goal of this study is for the recipients of a living related kidney transplant of one HLA haplotype to be withdrawn of immunosuppressive medication and become "tolerant "to their kidney graft. The recipient will receive a conditioning regimen composed of low dose radiation to the lymphoid tissue (total lymphoid irradiation, TLI) and anti-thymocyte globulin (ATG) at the time of transplant. They will then be infused with purified "stem cell" and T-cell from their kidney donors 2 weeks after the transplant to try to achieve mixed chimerism of their white blood cells with the donor (the recipient would have a mixture some of the with blood cells of the donor and theirs in their blood). The kidney donor has to provide peripheral stem cell 6-8 weeks before kidney donation. It is an outpatient procedure done using peripheral veins after treatment with G-CSF (filgrastim).Immunosuppressive medication will be decreased gradually and possibly stopped by 1 1/2 year after the transplantation if the recipient meets withdrawing criteria (persistence of mixed chimerism more than 18 months, no episode of rejection and no rejection on surveillance kidney biopsy). Potential candidates need to be approved for kidney transplant and available for close follow-up at Stanford University Medical Center.

ELIGIBILITY:
Inclusion Criteria:

1. All consenting adults who are 18 to 60 years, living donor transplant candidates and have a haplotype related living donor or > 2 HLA antigen matched, unrelated, living donor (including at least one HLA-DR antigen match plus at least one antigen match of either HLA-A or HLA-B).
2. Patients who agree to participate in the study and sign an Informed Consent.
3. Patients who have no known contraindication to administration of rabbit ATG or radiation.
4. Males and females of reproductive potential who agree to practice a reliable form of contraception for at least 24 months post-transplant.
5. ABO compatible.

Exclusion Criteria:

1. Previous treatment with rabbit ATG or a known allergy to rabbit proteins.
2. History of malignancy with the exception of non-melanoma skin malignancies.
3. Pregnant women or nursing mothers.
4. Serological evidence of HIV, Hepatitis B or Hepatitis C infection.
5. Seronegative for Epstein-Barr virus, if donor is seropositive.
6. Leukopenia (with a white blood cell count < 3000/mm3) or thrombocytopenia (with a platelet count < 100,000/mm3).
7. Panel Reactive Antibody greater than 80% or demonstration of donor specific antibody (DSA).
8. Prior organ transplantation.
9. High risk of primary kidney disease recurrence (e.g atypical HUS). However, patients with primary FSGS will not be excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2010-07-14 (Actual); Primary Completion 2024-06-14 (Estimated); Study Completion 2025-06-14 (Estimated)

PRIMARY OUTCOMES:
Long term freedom from transplant immunosuppressive drugs, safety, rate of infection, graft survival and patient survival. | 5 years and indefinitely if possible
  Subjects on study will have tapering of the immunosuppressive medication and withdrawal of the immunosuppressive medication if withdrawal criteria are met.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Busque, MD,MS, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Stanford University School of Medicine, Stanford, California
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scandling JD, Busque S, Dejbakhsh-Jones S, Benike C, Millan MT, Shizuru JA, Hoppe RT, Lowsky R, Engleman EG, Strober S. Tolerance and chimerism after renal and hematopoietic-cell transplantation. N Engl J Med. 2008 Jan 24;358(4):362-8. doi: 10.1056/NEJMoa074191. PMID 18216356
- [Background] Scandling JD, Busque S, Shizuru JA, Engleman EG, Strober S. Induced immune tolerance for kidney transplantation. N Engl J Med. 2011 Oct 6;365(14):1359-60. doi: 10.1056/NEJMc1107841. No abstract available. PMID 21991976
- [Background] Scandling JD, Busque S, Dejbakhsh-Jones S, Benike C, Sarwal M, Millan MT, Shizuru JA, Lowsky R, Engleman EG, Strober S. Tolerance and withdrawal of immunosuppressive drugs in patients given kidney and hematopoietic cell transplants. Am J Transplant. 2012 May;12(5):1133-45. doi: 10.1111/j.1600-6143.2012.03992.x. Epub 2012 Mar 8. PMID 22405058
- [Derived] Jensen KP, Hongo DA, Ji X, Zheng P, Pawar R, Wu TH, Busque S, Scandling JD, Shizuru JA, Lowsky R, Shori A, Dutt S, Waters J, Saraswathula A, Baker J, Tamaresis JS, Lavori P, Negrin R, Maecker H, Engleman EG, Meyer E, Strober S. Development of immunosuppressive myeloid cells to induce tolerance in solid organ and hematopoietic cell transplant recipients. Blood Adv. 2021 Sep 14;5(17):3290-3302. doi: 10.1182/bloodadvances.2020003669. PMID 34432869